CLINICAL TRIAL: NCT05443828
Title: Short-chain Fatty Acids in Plasma After Intake of Fermentable Cereal Fibres- An Extended Postprandial Study
Brief Title: Plasma SCFAs After Fermentable Cereal Fibres - A Postprandial Study
Acronym: FIFERM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, rivellese angela, Full Professor, Federico II University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 299/20
Record Dates: First submitted 2022-06-14; First posted 2022-07-05 (Actual); Last update posted 2022-07-05 (Actual); Status verified 2022-06

CONDITIONS: Overweight and Obesity
Keywords: dietary fiber; short chain fatty acids; butyrate; propionate; gut microbiota; glucose metabolism
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Extruded puff with vitacel (Active Comparator): The participants consumed a portion of extruded puff with added vitacel (cellulose) contained 11 g of fiber, in the context of a breakfast meal
  Interventions: Other: Breakfast Control Meal
- AX bread (Experimental): Participants consumed a portion of bread enriched with arabynoxylans (AX) contained 11 g of fiber, in the context of a breakfast meal
  Interventions: Other: Breakfast Test Meal
- Wheat bran puff (Experimental): Participants consumed a portion of wheat bran puff contained 11 g of fiber, in the context of a breakfast meal
  Interventions: Other: Breakfast Test Meal

INTERVENTIONS:
Other: Breakfast Control Meal — The participants consumed extruded puff with added vitacel (cellulose) as part of the breakfast meal (400 kcal, 12 g fiber) followed by consumption of standardised meal at lunch and dinner . The lunch and dinner did noft contain any intervention products. Blood samples were collected at 14 timepoints drawn (first sample 15 minutes before breakfast, last sample 24 hours after breakfast), during 6 hours after the test breakfast meal and during other 2 hours after standardised lunch.
  Other Names: Breakfast Meal with vitacel puff
  Arms: Extruded puff with vitacel
Other: Breakfast Test Meal — The participants consumed bread with added arabynoxylans (AX) as part of the breakfast meal (400 kcal, 12 g fiber) followed by consumption of standardised meal at lunch and dinner . The lunch and dinner did noft contain any intervention products. Blood samples were collected at 14 timepoints drawn (first sample 15 minutes before breakfast, last sample 24 hours after breakfast), during 6 hours after the test breakfast meal and during other 2 hours after standardised lunch.
  Other Names: Breakfast Meal with AX bread
  Arms: AX bread
Other: Breakfast Test Meal — The participants consumed extruded puff with added wheat bran as part of the breakfast meal (400 kcal, 12 g fiber) followed by consumption of standardised meal at lunch and dinner . The lunch and dinner did noft contain any intervention products. Blood samples were collected at 14 timepoints drawn (first sample 15 minutes before breakfast, last sample 24 hours after breakfast), during 6 hours after the test breakfast meal and during other 2 hours after standardised lunch.
  Other Names: Breakfast Meal with extruded puff with added wheat bran
  Arms: Wheat bran puff

SUMMARY:
Circulating SCFAs reflect the net effect of what is produced in the large intestine from dietary fibre fermentation, bioavailability after considerable absorption by the enterocytes and in the liver and the elimination. It is yet unclear to what extent SCFA levels in systemic circulation is of importance for metabolic disease risk and diabetes aetiology. Recent high-impact studies strongly suggest beneficial metabolic effects of butyrate and adverse effects from propionate However, no study has yet investigated to what extent butyrate or propionate producing diets may influence metabolic risk factors for T2D across individuals with different butyrate or propionate producing capacity. The overall aim is to investigate individual's ability to generate high concentrations of butyrate and propionate in plasma after acute intake of different fibre rich foods in an extended postprandial setting. The aim is further to optimize time points for data collection to allow robust assessment of plasma-time concentration profiles of butyrate and propionate to establish a screening approach to identify individuals with high/low butyrate/propionate plasma concentrations. This will be used in later precision nutrition studies where diet will be tailored to high/low SCFA-metabotypes.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) 20-35 kg/m2
* Waist circumference >102 cm (males) or 88 cm (females)
* Haemoglobin, low density lipoprotein (LDL) cholesterol or triglycerides within the normal reference ranges (age and sex specific) according to the laboratory analysing the screening samples.
* Willing to collect faecal samples at home and store them in their household freezer

Exclusion Criteria:

* Blood donation or participation in a clinical study with blood sampling within 30 days prior to screening visit and throughout the study
* Having been treated with antibiotics within the past 3 months or planning to undergo treatment during the study period.
* Diastolic blood pressure ³ 105 mm Hg at visit 1
* Systolic blood pressure ³ 160 mm at visit 1
* History of stomach or gastrointestinal conditions (Inflammatory bowel disease, Crohn's disease, malabsorption etc.)
* More than 10 hours physical activity per week
* History of heart failure or heart attack within 1 year prior to screening
* Having type I and type 2 diabetes
* Previous gastrointestinal surgery (e.g., gastric bypass, gastric sleeve, bowel resection, colostomy etc.), with the exception of minor surgeries such removal of appendix or gall bladder at least 6 months prior to screening.
* Thyroid disorder not controlled by drug therapy
* History of drug or alcohol abuse
* Stroke or transient ischemic attack (TIA) within 1 year prior to screening
* Consumption of drugs aimed at weight management or drugs affecting body weight to a degree that is considered unsuitable for study participation by responsible physician.
* Pregnant, lactation or planning a pregnancy within the timeframe of the study. Pregnancy must have ended at least 6 months prior to screening, and lactation must have ended at least 1 month prior to screening.
* Food allergies or intolerances preventing consumption of any products included in the study
* Strict vegetarian/vegan (participants must be able to consume the standardized meals used in the study)

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2021-11-09 (Actual); Primary Completion 2022-05-24 (Actual); Study Completion 2022-05-24 (Actual)

PRIMARY OUTCOMES:
Differences in plasma propionate and butyrate concentration | 24 hours
  Differences in plasma SCFA concentration- time profiles , with emphasis on butyrate and propionate concentrations after intake of the breakfast meals cointaned the same amount of different fibre sources (wheat bran puff and Arabynoxylans bread) compared to control fiber (extruded vitacel puff). Plasma SCFAs concentration was evaluated by LC-MS analysis

SECONDARY OUTCOMES:
Effects of the different fibres sources on plasma glucose | 24 hours
  Differences in postprandial plasma glucose concentrations after intake of the breakfast meals cointaned the same amount of different fibre sources (wheat bran puff and Arabynoxylans bread) compared to control fiber (extruded vitacel puff). Plasma glucose concentration was measured by enzymatic colorimetric methods
Effects of the different fibres sources on plasma insulin | 24 hours
  Differences in postprandial plasma insulin concentrations after intake of the breakfast meals cointaned the same amount of different fibre sources (wheat bran puff and Arabynoxylans bread) compared to control fiber (extruded vitacel puff). Plasma insulin concentration was measured by ELISA method
Effects of the different fibres sources on plasma free fatty acids | 24 hours
  Differences in postprandial plasma free fatty acids (FFA) concentrations after intake of the breakfast meals cointaned the same amount of different fibre sources (wheat bran puff and Arabynoxylans bread) compared to control fiber (extruded vitacel puff). Plasma FFA concentration was measured by enzymatic colorimetric method
Effects of the different fibres sources on plasma GLP-1 | 24 hours
  Differences in postprandial plasma glucagon like peptide 1 (GLP1) concentrations after intake of the breakfast meals cointaned the same amount of different fibre sources (wheat bran puff and Arabynoxylans bread) compared to control fiber (extruded vitacel puff). Plasma GLP1 concentration was measured by ELISA method
Gut microbiota composition | 24 hours
  Analysis of the gut microbiota composition from faecal samples collected at fasting before the intake of the breakfast meals cointaned the same amount of different fibre sources (wheat bran puff and Arabynoxylans bread) compared to control fiber (extruded vitacel puff). Faecal microbiota composition was evaluated by 16S rRNA sequencing.

CONTACTS AND LOCATIONS:
Overall Officials: Angela Rivellese, MD, Study Chair — Federico II University
Locations (1):
- Department of Clinical Medicine and Surgery Federico II University, Naples, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Baxter NT, Schmidt AW, Venkataraman A, Kim KS, Waldron C, Schmidt TM. Dynamics of Human Gut Microbiota and Short-Chain Fatty Acids in Response to Dietary Interventions with Three Fermentable Fibers. mBio. 2019 Jan 29;10(1):e02566-18. doi: 10.1128/mBio.02566-18. PMID 30696735
- [Result] Chambers ES, Preston T, Frost G, Morrison DJ. Role of Gut Microbiota-Generated Short-Chain Fatty Acids in Metabolic and Cardiovascular Health. Curr Nutr Rep. 2018 Dec;7(4):198-206. doi: 10.1007/s13668-018-0248-8. PMID 30264354
- [Result] Kim CH. Microbiota or short-chain fatty acids: which regulates diabetes? Cell Mol Immunol. 2018 Feb;15(2):88-91. doi: 10.1038/cmi.2017.57. Epub 2017 Jul 17. No abstract available. PMID 28713163
- [Result] Kovatcheva-Datchary P, Nilsson A, Akrami R, Lee YS, De Vadder F, Arora T, Hallen A, Martens E, Bjorck I, Backhed F. Dietary Fiber-Induced Improvement in Glucose Metabolism Is Associated with Increased Abundance of Prevotella. Cell Metab. 2015 Dec 1;22(6):971-82. doi: 10.1016/j.cmet.2015.10.001. Epub 2015 Nov 6. PMID 26552345
- [Derived] Costabile G, Vitale M, Testa R, Rivieccio A, Palmnas M, Lopez-Sanchez P, Landberg R, Riccardi G, Giacco R. Daily profiles of plasma short-chain fatty acids after the intake of three different cereal fibers: a randomized controlled study. Eur J Nutr. 2025 Jun 11;64(5):217. doi: 10.1007/s00394-025-03741-7. PMID 40498116